CLINICAL TRIAL: NCT04175210
Title: Prospective Randomized Study of Accelerated Radiation Therapy (PRART) : A Non-Inferiority Trial to Compare Breast Cosmesis and Local Control After Concomitant Boost Breast Radiotherapy With Fifteen Fractions in Three Weeks (Arm 1, Standard) Versus Ten Fractions in Two Weeks (Arm 2, Experimental)
Brief Title: Prospective Randomized Study of Accelerated Radiation Therapy (PRART)
Acronym: PRART
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-07020533
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARM 1-4050cGY and boost to tumor bed of 4800cGY in 15fractions (Experimental): Patients randomized to ARM 1 will receive whole breast radiotherapy of 4050cGY and a concomitant boost to the tumor bed of 4800cGY in 15 fractions
  Interventions: Radiation: Radiation therapy - 3 weeks
- ARM 2 - 3200cGY and boost to tumor bed of 4200cGY -10fractions (Experimental): Patients randomized to ARM 2 will receive whole breast radiotherapy of 3200cGY and a concomitant boost to the tumor bed of 4200cGY in 10 fractions.
  Interventions: Radiation: Radiation therapy - 2 weeks

INTERVENTIONS:
Radiation: Radiation therapy - 3 weeks — Patients randomized to ARM 1 will receive whole breast radiotherapy of 4050cGY and a concomitant boost to the tumor bed of 4800cGY in 15 fractions
  Arms: ARM 1-4050cGY and boost to tumor bed of 4800cGY in 15fractions
Radiation: Radiation therapy - 2 weeks — Patients randomized to ARM 2 will receive whole breast radiotherapy of 3200cGY and a concomitant boost to the tumor bed of 4200cGY in 10 fractions.
  Arms: ARM 2 - 3200cGY and boost to tumor bed of 4200cGY -10fractions

SUMMARY:
Patients with Stage 0 ductal carcinoma in situ (Tis (DCIS), Stage T1-T2, lymph node negative(N0) breast cancers will be randomized to receive whole breast radiotherapy with a concomitant boost to the tumor bed over 15 fractions (Arm 1, standard) versus 10 fractions (Arm 2, experimental).

ELIGIBILITY:
Inclusion Criteria:

* Women status post segmental mastectomy
* If unilateral, pT1-2 breast cancer excised with negative margins
* If bilateral, pT1-2 breast cancer excised with negative margins AND/OR pTis excised with negative margins.
* Clinically N0 or pN0 or sentinel node negative
* Ductal carcinoma in situ DCIS with negative margins (no DCIS on inked margins).
* Women with previous contralateral breast cancer.

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast.
* 90 days from last surgery, unless s/p adjuvant chemotherapy
* 60 days from last chemotherapy
* Male breast cancer

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with acute toxicity grade ≥ 2 on the 10-fraction arm compared to proportion of patients with acute toxicity grade ≥ 2 on the 15-fraction arm evaluated up to 1-month post-radiation treatment | up to 1-month post-radiation treatment
  Rate of grade ≥ 2 of acute toxicity defined according to the Common Terminology Criteria for Adverse Events (CTCAEs) - version 5.0, on the 10-fraction arm compared to the rate on the 15-fraction arm will be measured, up to 1-month post-radiation treatment.

SECONDARY OUTCOMES:
Proportion of patients with local breast cancer control on the 10-fraction arm compared to proportion of patients with local breast cancer control on the 15-fraction arm evaluated at 2-3 years post-radiation treatment | 2-3 years
  Assess and compare local control at 2-3 years between the two arms. At each post treatment follow-up visit, a physical exam to detect breast clinical recurrence will be performed. Mammographic studies and/or breast MRI will be performed and reviewed on an annual basis, according to the standard care. Local control will be defined according to the findings from physical exam, mammographic studies and/or breast MRI.
Proportion of patients with local breast cancer control on the 10-fraction arm compared to proportion of patients with local breast cancer control on the 15-fraction arm evaluated at 5 years post-radiation treatment | 5 years
  Assess and compare local control at 5 years between the two arms. At each post treatment follow-up visit, a physical exam to detect breasts clinical disease recurrence will be performed. Mammographic studies and/or breast MRI will be performed and reviewed on an annual basis, according to the standard care. Local control will be defined according to the findings from physical exam, mammographic studies and/or breasts MRI.
Number of subjects with fibrosis defined per grades according to LENT/SOMA fibrosis scoring system on the 10-fraction arm and on the 15-fraction arm evaluated at 2-3 years post-radiation treatment | 2-3 years
  Assess and compare fibrosis at 2-3 years between the two arms. At each post treatment follow-up visit, the fibrosis will be assessed by breasts palpation performed by the physician or nurse practitioner and will be measured as per LENT/SOMA fibrosis scoring system. According to this scoring system, fibrosis is categorized into three grades (Grade 1, Grade 2 and Grade 3), where Grade 1 is defined as "barely palpable, increased density" and Grade 3 is defined as "very marked density, retraction, and fixation".
Number of subjects reporting breast cosmesis according to BCTOS questionnaire on the 10-fraction arm and on the 15-fraction arm evaluated at 2-3 years post-radiation treatment | 2-3 years
  Assess and compare breast cosmesis at 2-3 years between the two arms. At each post treatment follow-up visit, breast cosmesis will be self-assessed by the patient using Breast Cancer Treatment Outcome Scale (BCTOS) questionnaires. According to this scale, breast cosmesis is evaluated using a four-point system (Point 1, Point 2, Point 3, and Point 4), where Point 1 is defined as "no change compared to the untreated breast" and Point 4 as "large change compared to the untreated breast."
Number of subjects with fibrosis defined per grades according to LENT/SOMA fibrosis scoring system on the 10-fraction arm and on the 15-fraction arm evaluated at 5 years post-radiation treatment | 5 years
  Assess and compare fibrosis at 5 years between the two arms. At each post treatment follow-up visit, the fibrosis will be assessed by breasts palpation performed by the physician or nurse practitioner and will be measured as per LENT/SOMA fibrosis scoring system. According to this scoring system, fibrosis is categorized into three grades (Grade 1, Grade 2 and Grade 3), where Grade 1 is defined as "barely palpable, increased density" and Grade 3 is defined as "very marked density, retraction, and fixation".
Number of subjects reporting breast cosmesis according to BCTOS questionnaire on the 10-fraction arm and on the 15-fraction arm evaluated at 5 years post-radiation treatment | 5 years
  Assess and compare breast cosmesis at 5 years between the two arms. At each post treatment follow-up visit, breast cosmesis will be self-assessed by the patient using Breast Cancer Treatment Outcome Scale (BCTOS) questionnaires. According to this scale, breast cosmesis is evaluated using a four-point system (Point 1, Point 2, Point 3, and Point 4), where Point 1 is defined as "no change compared to the untreated breast" and Point 4 as "large change compared to the untreated breast."

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - New York Presbyterian Hospital at Lower Manhattan Cancer Center, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No